CLINICAL TRIAL: NCT03359174
Title: An Efficacy Trial of Low Dose All-trans Retinoic Acid (ATRA) in Patients With Primary Sclerosing Cholangitis
Brief Title: An Efficacy Trial of Low Dose All-trans Retinoic Acid in Patients With Primary Sclerosing Cholangitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000021447
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Cholangitis, Sclerosing
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All-trans retinoic acid (ATRA) therapy (Experimental): Fixed low dose of ATRA 10 mg twice daily for 24 weeks.
  Interventions: Drug: All-trans retinoic acid

INTERVENTIONS:
Drug: All-trans retinoic acid — Fixed low dose of ATRA 10 mg twice daily for 24 weeks.

SUMMARY:
The purpose of this research study is to determine whether a low dose of ATRA will improve laboratory tests of liver and bile duct inflammation in patients with PSC. The investigators will also look for changes to other blood tests which are related to inflammation, scarring, and the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18-80
* Diagnosis of large-duct PSC based on ERCP or MRCP, or liver biopsy findings without alternative explanation for findings, for at least 6 months.
* Serum ALP levels persistently more than 1.5 x upper limit of normal over the past 6 months.
* Ursodeoxycholic acid therapy must be discontinued for at least 3 months.
* At least 2 forms of barrier protection for males and females of child-bearing age.

Exclusion Criteria:

* Small duct PSC, overlap with autoimmune hepatitis, IgG4 disease or secondary sclerosing cholangitis.
* Any malignancy, presently or within the past 5 years, except adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix or in situ prostate cancer.
* Viral hepatitis including hepatitis A, B, C, D, E.
* Decompensated cirrhosis, or planned liver transplantation.
* Recent diagnostic or therapeutic biliary manipulation (endoscopic, radiologic) within the past 3 months.
* Ascending Cholangitis requiring antibiotics within the past 3 months.
* Uncontrolled IBD, or IBD requiring the use of steroids.
* Acute or Chronic Kidney Disease with serum creatinine > 2 mg/dL.
* Allergy to ATRA or vitamin A compounds.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Boyer, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from physicians case load at Yale University, Digestive Disease's Liver clinic between May 2018 and December 2018. Both participants were enrolled in May of 2018.
Pre-assignment Details: Of the two patients who screened, both met inclusion and exclusion criterial and were enrolled
Period: Overall Study
Arm/Group | All-trans Retinoic Acid (ATRA) Therapy
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | All-trans Retinoic Acid (ATRA) Therapy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change of Serum Alkaline Phosphatase (ALP)
Description: Blood will be drawn at each time point to compare pre- and post-treatment values for each individual.
Time Frame: Baseline to week 24.
Population: Data were not collected
Arm/Group | All-trans Retinoic Acid (ATRA) Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Patients Who Have Normalization of Serum ALP or Reduction to Less Than 1.5 x Upper Limit of Normal (ULN)
Description: Blood is drawn at each time point to assess the outcome.
Time Frame: Baseline to week 24.
Population: Only 1 patient completed the study, and no trial end point was achieved so there was no data to record. .
Arm/Group | All-trans Retinoic Acid (ATRA) Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: The Percent of Patients Who Have Reduction of Serum C4 by 50%
Description: Blood is drawn at each time point to assess the outcome.
Time Frame: Baseline to week 24.
Population: Only 1 patient completed the study, data not reported.
Arm/Group | All-trans Retinoic Acid (ATRA) Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: The Percent of Patients Who Have Reduction of Serum Bile Acids by 50%
Description: Blood is drawn at each time point to assess the outcome.
Time Frame: Baseline to week 24.
Population: Only 1 patient completed the study, data not reported.
Arm/Group | All-trans Retinoic Acid (ATRA) Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: The Percent of Patients Who Have Reduction of Serum Alanine Aminotransferase (ALT) by 50%
Description: Blood is drawn at each time point to assess the outcome.
Time Frame: Baseline to week 24.
Population: Only 1 patient completed the study, data not reported.
Arm/Group | All-trans Retinoic Acid (ATRA) Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: The Percent of Patients Who Have Reduction of Serum Enhanced Liver Fibrosis Score (ELF) by 10%
Description: Blood is drawn at each time point to assess the outcome.
Time Frame: Baseline to week 24.
Population: Only 1 patient completed the study, data not reported.
Arm/Group | All-trans Retinoic Acid (ATRA) Therapy
Number analyzed (Participants) | 0

7. Secondary Outcome: The Percent of Patients Who Have Improvement in Fibrosis Per Transient Elastography by at Least 1 Stage
Description: Transient Elastography will be performed at baseline and week 24 to assess the outcome.
Time Frame: Baseline to week 24.
Population: Only 1 patient completed the study, data not reported.
Arm/Group | All-trans Retinoic Acid (ATRA) Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 28 weeks post treatment initiation.
Arm/Group | All-trans Retinoic Acid (ATRA) Therapy
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All-trans Retinoic Acid (ATRA) Therapy (N=2)
alkaline phosphatase increase (Hepatobiliary disorders) | 1 (1)
Blood bilirubin increased (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT03359174/Prot_SAP_000.pdf